CLINICAL TRIAL: NCT04563832
Title: Self-administered Hyperinsufflation Chest Mobilization Randomized Study on the Risk of Low Respiratory Infection in Patients With Multiple Sclerosis With Sputum Capacity Deficit
Brief Title: Self-administered Hyperinsufflation Chest on the Risk of Low Respiratory Infection in Patients With Multiple Sclerosis With Sputum Capacity Deficit
Acronym: MS-COUGH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP2020
Record Dates: First submitted 2020-09-21; First posted 2020-09-24 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2021-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: * Control group: standardized respiratory management.
  * Experimental group: same program, associated with the daily use of a hyperinsufflation technique.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): standardized respiratory management.
  Interventions: Other: Standardized respiratory management program
- Experimental group (Experimental): same program as control group associated with the daily use of a hyperinsufflation technique (2 times per day during15 minutes, 5 days a week, for 2 years)
  Interventions: Other: Standardized respiratory management program; Other: CoughAssist

INTERVENTIONS:
Other: Standardized respiratory management program — Bronchial decluttering education, respiratory physiotherapy, specialized medical follow-up for 2 years
Other: CoughAssist — self-administered mechanical in-exsufflation - CoughAssist (2 x 15 min per day, 5 days per week for 2 years)
  Arms: Experimental group

SUMMARY:
In patients with neuromuscular disease, chest mobilization by hyperinsufflation slows respiratory decline by almost 80% compared to controls, and prevents complications like pneumonia, atelectasis and respiratory distress.

This insufflation technique improves the airway clearance and reduces the need for invasive ventilation. It also improves CV and DEPtoux in patients with neuromuscular pathology

DETAILED DESCRIPTION:
During multiple sclerosis (MS), although expiratory involvement and reduced sputum capacity are predominant, automated techniques of hyperinsufflation and in-exsufflation remain underused and undervalued. A single retrospective study suggests a decrease in the decline in respiratory function with regular manual hyperinsufflation.

Evidence of a benefit of chest mobilization by hyperinsufflation by a controlled trial is therefore necessary before recommending its use in MS.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed MS diagnosis (McDonald criteria)
* EDSS ≥ 7
* Age greater than or equal to 18 years.
* Expiratory flow during a coughing effort (DEPtoux) ˂4.5L / s.

Exclusion Criteria:

* ENT and / or thoracic surgery less than 6 months old
* Progressive or past pneumothorax / pneumomediastinum
* Severe swallowing disorders.
* Inability to use the device under study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-11-25 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of a self-administered automated hyperinsufflation technique for 2 years, versus standard management, on respiratory infection risk within 2 years after randomization, in patients with MS. | 24 months
  This will be evaluated by the incidence of lower respiratory infections requiring antibiotic therapy

SECONDARY OUTCOMES:
Effect of COUGH-ASSIST on slowing the decline in respiratory function, | 12 months and 24 months
  This will be demonstrated by monitoring respiratory function by spirometry
Functional effectiveness of COUGH-ASSIST | 12 months and 24 months
  By using the goal attainmentscaling method (GAS)
Tolerance and compliance with COUGH-ASSIST, | 24 months
  This will be evaluated via an online "patient reported outcomes form" and data readings from the internal memory of the COUGH-ASSIST
Effectiveness of COUGH-ASSIST in reducing the risk of serious respiratory infection | 24 months
  This will be evaluate by the number of serious respiratory infection

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Raymond Poincaré, Garches, Haut de Seine, France